CLINICAL TRIAL: NCT00439413
Title: Phase 2, Double-Blind, Placebo-Controlled Trial of Selegiline Transdermal System (STS) as an Aid for Smoking Cessation.
Brief Title: Selegiline for Smoking Cessation - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIDA-CSP-1022-1; NCT00462514 (obsolete NCT alias)
Record Dates: First submitted 2007-02-22; First posted 2007-02-23 (Estimated); Results first posted 2016-10-13 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Selegiline Transdermal Patch (Active Comparator): Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -4 week Screening/Baseline Phase.
  During treatment, subjects received Selegiline Transdermal System, 6mg -20cm(2) patch, one time per day for 9 weeks
  Subjects were provided with on-site, individual smoking cessation counseling sessions 1x per week for 9 weeks
  Interventions: Drug: Selegiline Transdermal Patch; Behavioral: Smoking Cessation Counseling
- Placebo (Placebo Comparator): Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during a -4 week Screening/Baseline Phase.
  During treatment, subjects received matched placebo 20cm(2) patch transdermal patch one time per day for 9 weeks
  Subjects were provided with on-site, individual smoking cessation counseling sessions 1x per week for 9 weeks
  Interventions: Drug: Placebo; Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Drug: Selegiline Transdermal Patch — Selegiline cm(2) via transdermal system
  Other Names: STS Patch
  Arms: Selegiline Transdermal Patch
Drug: Placebo — Matching placebo via transdermal system
  Other Names: Placebo Patch
  Arms: Placebo
Behavioral: Smoking Cessation Counseling — Subjects were provided with on-site, individual smoking cessation counseling sessions 1x per week for 9 weeks

SUMMARY:
The purpose of this study is designed to examine the effects of Selegiline Transdermal System and behavioral intervention in smoking cessation as compared to behavioral intervention alone.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age
* Be in good general health
* Must meet Diagnostic and Statistical Manual-IV (DSM-IV) diagnostic criteria for nicotine dependence
* Be currently smoking > 15 cigarettes/day, and have smoked cigarettes for the past 5 years
* Subjects must be motivated to quite smoking
* If female and of child bearing potential, agrees to use birth control and subject
* Subject must be able to understand and provide written informed consent.

Exclusion

Criteria:

* Please contact site for more information

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2007-06; Primary Completion 2008-08 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elbert D Glover, Ph.D., Principal Investigator — VA Medical Center
Locations (4):
- United States (4):
  - Department of Public & Community Health, College Park, Maryland
  - Robert Wood Johnson Med School-Tobacco Dep Program, New Brunswick, New Jersey
  - Tri-State Tobacco and Alcohol Research Center, Cincinnati, Ohio
  - Center For Tobacco Research and Intervention, Milwaukee, Wisconsin

REFERENCES:
- [Result] Kahn R, Gorgon L, Jones K, McSherry F, Glover ED, Anthenelli RM, Jackson T, Williams J, Murtaugh C, Montoya I, Yu E, Elkashef A. Selegiline transdermal system (STS) as an aid for smoking cessation. Nicotine Tob Res. 2012 Mar;14(3):377-82. doi: 10.1093/ntr/ntr143. Epub 2011 Aug 16. PMID 21846661
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Groups:
- Selegiline Transdermal System: Participants received Selegiline Transdermal System (STS) 20 mg x 20 cm patch applied daily for 10 weeks
- Placebo: Participants received Selegiline Transdermal System (STS) 20 mg x 20 cm placebo patch applied daily for 10 weeks
Period: Overall Study
Arm/Group | Selegiline Transdermal System | Placebo
Started | 121 | 125
Completed | 90 | 88
Not Completed | 31 | 37

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Selegiline Transdermal System | Placebo | Total
Number analyzed (Participants) | 121 | 125 | 246
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (14.2) | 47.3 (13.6) | 46.5 (14)
Gender [Count of Participants; unit: Participants]
  Female | 62 | 59 | 121
  Male | 59 | 66 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 6 | 5 | 11
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 30 | 59
  White | 86 | 87 | 173
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 121 | 125 | 246

OUTCOME MEASURES:

1. Primary Outcome: Quit Rate
Description: The number of subjects in each treatment group who ceased smoking as measured by four weeks of self-reported abstinence confirmed by at least two exhales - carbon monoxide (CO) measurements during the last four weeks of treatment (study weeks 6 through 9).
Time Frame: Study weeks 6 through 9
Measure: Number; unit: participants
Groups:
- Selegiline Transdermal System: Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during -2 to -1 week Screening/Baseline Phase.
  During treatment, subjects received 20mg x 20cm Selegiline Transdermal System patch, once daily for 10 weeks.
  Subjects were provided on-site brief counseling sessions 1x per week for 9 weeks.
- Matching Placebo: Subjects were evaluated for their compliance with protocol inclusion/exclusion criteria during -2 to -1 week Screening/Baseline Phase.
  During treatment, subjects received 20mg x 20cm Selegiline Transdermal System placebo patch, once daily for 10 weeks.
  Subjects were provided on-site brief counseling sessions 1x per week for 9 weeks.
Arm/Group | Selegiline Transdermal System | Matching Placebo
Number analyzed (Participants) | 121 | 125
participants | 18 | 15

2. Secondary Outcome: Abstinence
Description: The proportion is determined by dividing the number who achieved abstinence at the end of treatment as defined for the primary outcome measure and are still abstinent by self report and separately by self report with confirmation by exhaled CO by the total number randomized to the treatment group.
Time Frame: week 14
Measure: Number; unit: participants
Arm/Group | Selegiline Transdermal System | Placebo
Number analyzed (Participants) | 121 | 125
participants | 16 | 10

ADVERSE EVENTS:
Time Frame: Week 2 through 9 and follow-up weeks (10 and 14)
Arm/Group | Selegiline Transdermal System | Matching Placebo
Serious Adverse Events (participants affected / at risk) | 3/121 | 0/125
Other Adverse Events (participants affected / at risk) | 99/121 | 76/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selegiline Transdermal System (N=121) | Matching Placebo (N=125)
Fracture of femur (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Heart Attack (Cardiac disorders) | 1 (1) | 0 (0)
Exacerbation of COPD dut to pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selegiline Transdermal System (N=121) | Matching Placebo (N=125)
Headache (Nervous system disorders) | 18 (23) | 24 (35)
Application Site Erythema (General disorders) | 13 (14) | 4 (4)
Dry Mouth (Gastrointestinal disorders) | 9 (9) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 8 (9)
Insomnia (Psychiatric disorders) | 19 (19) | 10 (12)
Nasopharyngitis (Infections and infestations) | 6 (7) | 7 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (5)
Skin irritation (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (5)
Blood pressure increased (Investigations) | 1 (2) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 1 (1)
Tooth extraction (Surgical and medical procedures) | 4 (4) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 2 (2)
Vision blurred (Eye disorders) | 2 (2) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Hypersensitivity (Hepatobiliary disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days